CLINICAL TRIAL: NCT05412888
Title: The Effect of Ischemic Preconditioning and Physical Exercise on the Endocrine Function of Skeletal Muscle - the Effect of CoQ10 Supplementation. In Vivo and in Vitro Studies.
Brief Title: Effect of CoQ10 on the Endocrine Function of Skeletal Muscle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MUGdansk CoQ10
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Ischemic Preconditioning; Coenzyme Q Deficiency; Exercise Training
Keywords: skeletal muscle; myokines; ischemia; inflammation
MeSH Terms: conditions — Coenzyme Q10 Deficiency; Ischemia; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supplemented population 300mg (Placebo Comparator): Supplemented population 300mg/24h CoQ10 - 25 participants
  Interventions: Dietary Supplement: CoQ10 supplementation
- Training and IPC preconditioning (Experimental): Group subjected to training and preconditioning by ischemia (IPC training) - 25 participants,
  Interventions: Procedure: Ischemic preconditioning training
- Control group (placebo) (Placebo Comparator): Control group to CoQ10 supplementation (placebo)- 25 participants
  Interventions: Dietary Supplement: Sham IPC combined with placebo
- IPC control group (Sham Comparator): IPC control group - 25 participants
  Interventions: Dietary Supplement: IPC training combined with CoQ10 supplementation

INTERVENTIONS:
Dietary Supplement: CoQ10 supplementation — Young men training endurance running will be supplemented with CoQ10
  Arms: Supplemented population 300mg
Procedure: Ischemic preconditioning training — Young men training endurance running will undergo IPC training
  Arms: Training and IPC preconditioning
Dietary Supplement: IPC training combined with CoQ10 supplementation — Young men training endurance running will undergo IPC training combined with CoQ10 supplementation
  Arms: IPC control group
Dietary Supplement: Sham IPC combined with placebo — Young men training endurance running will undergo sham IPC training combined with placebo supplementation
  Arms: Control group (placebo)

SUMMARY:
Recent studies have also shown that repeated episodes of ischemia, followed by reperfusion (IPC), can contribute to the development of adaptive changes not only in the area of the heart muscle, but also in the structure of the skeletal muscles.

In the project, several research questions will be evaluated e.g. what is the relationship between oxidative stress parameters, uric acid concentration and nitric oxide degradation products in groups of people undergoing two-week training in ischemic training, or what is the relationship between the expression of genes associated with muscle cell growth (e.g. myostatin gene) and the effect of ischemia preconditioning training etc.

DETAILED DESCRIPTION:
Both in sport and medicine, methods are constantly sought that can significantly contribute to improving the ability of tissues to perform their functions and protecting them from effort-induced damage.

In a wide range of interests, especially in people treated for ischemic changes of cardiovascular diseases, are protocols of tissue preconditioning by transient ischemia which significantly contribute to the increase in blood flow in tissue structure.

Recent studies have also shown that repeated episodes of ischemia, followed by reperfusion (IPC), can contribute to the development of adaptive changes not only in the area of the heart muscle, but also in the structure of the skeletal muscles. There is still a lack of detailed research on genetic conditions related to adaptive changes in this area of interest.

In the project, the following research questions were posed:

1. What is the relationship between oxidative stress parameters, uric acid concentration and nitric oxide degradation products in groups of people undergoing two-week training in IPC training, or 2 weeks of CoQ10 supplementation in the light of non-training and non-supplementation?
2. What is the relationship between two weeks of lower limb ischemia preconditioning training, or CoQ10 supplementation, and the expression of genes associated with the stress response (HSF-1, NF-kB, TNF dependent glass)?
3. What is the relationship between the expression of genes associated with muscle cell growth (e.g. myostatin gene) and the effect of preconditioning training by ischemia?
4. What is the relationship between the expression of genes associated with intracellular metabolism and the effect of CoQ10 supplementation?
5. What is the relationship between the expression of genes encoding enzymes of energy pathways (e.g. GAPDH, LDH) and IPC training or CoQ10 supplementation in the study group?
6. How does IPC training or CoQ10 supplementation affect the expression of genes responsible for membrane transport, and the Hedgehog pathway in muscle cells (including Gli1)?
7. How does IPC training affect the expression of transcription factors: Hif-1-alpha (hypoxia-induced factor) and NF-kB and selected genes dependent on their activity?

HYPOTHESIS The level of gene expression associated with oxidative stress, muscle fiber development, angiogenesis, muscle cell energy, and membrane transport will change under the influence of the use of preconditioning training by deficiency or CoQ10 supplementation

ELIGIBILITY:
Inclusion Criteria: - gender (males only),

* not taking medication during the study,
* good health (no concomitant injuries),
* negative history of cardiovascular disorders, autonomic nervous system, mental disorders, cerebrospinal injuries and other diseases that may directly affect the results obtained.

Exclusion Criteria:

Lack of consent to participate in the research project or negative result of medical examinations.

Ages: 21 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The effects of IPC on physical performance | 8 weeks
  IPC training will be combined with endurance exercise and VO2max and serum Lactate will be measured
The effects of CoQ10 supplementation on physical performance | 8 weeks
  CoQ10 supplementation combined with endurance training will be evaluated for endurance improvement in young men. VO2max, myokines, genes associated with the stress response will be measured
The effects of CoQ10 supplementation and IPC on physical performance | 8 weeks
  CoQ10 supplementation combined with IPC and endurance training will be evaluated for endurance improvement in young men. VO2max, myokines, genes associated with the stress response, ulic acid will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Jedrzej Antosiewicz, Gdansk, Pomeranian Voivodeship, Poland